CLINICAL TRIAL: NCT02370537
Title: A Two-part, Open-label, Randomised, Crossover, Multicentre, Phase II Study to Investigate the Presence of Pancreatic Exocrine Insufficiency (PEI) in Patients With Type 2 Diabetes Mellitus, and to Investigate the Pharmacokinetics of EPANOVA® and OMACOR® Following a Single Oral Dose in Patients With Different Degrees of PEI
Brief Title: A Study to Investigate How Common Pancreatic Exocrine Insufficiency (PEI) is in Patients With Type 2 Diabetes and Also to Investigate the Uptake of a Single Dose of EPANOVA® or OMACOR® in Patients With Different Degrees of PEI
Acronym: PRECISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5881C00006; 2014-003511-11 (EudraCT Number)
Record Dates: First submitted 2015-02-24; First posted 2015-02-25 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2; Exocrine Pancreatic Insufficiency
Keywords: omega-3 carboxylic acid
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Exocrine Pancreatic Insufficiency | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence AB (Experimental): A single dose of EPANOVA® 4 g (administered as 4 x 1 g capsules) at Visit 4, followed by 10 to 14 days washout, followed by a single dose of OMACOR® 4 g (administered as 4 x 1 g capsules) at Visit 7.
  Interventions: Drug: Epanova® (omega-3 carboxylic acids); Drug: Omacor® (omega-3-acid ethyl esters)
- Sequence BA (Experimental): A single dose of OMACOR® 4 g (administered as 4 x 1 g capsules) at Visit 4, followed by 10 to 14 days washout, followed by a single dose of EPANOVA® 4 g (administered as 4 x 1 g capsules) at Visit 7.
  Interventions: Drug: Epanova® (omega-3 carboxylic acids); Drug: Omacor® (omega-3-acid ethyl esters)

INTERVENTIONS:
Drug: Epanova® (omega-3 carboxylic acids) — 4 g (administered orally as 4 x 1 g capsules)
  Other Names: omega-3 carboxylic acids
Drug: Omacor® (omega-3-acid ethyl esters) — 4 g (administered orally as 4 x 1 g capsules)
  Other Names: omega-3-acid ethyl esters

SUMMARY:
This study is a 2-part open-label, randomized, crossover, multicenter, non-therapeutic Phase II study to investigate the presence of pancreatic exocrine insufficiency (PEI) in patients with Type 2 diabetes mellitus (T2DM), and to investigate the pharmacokinetics (PK) of EPANOVA® (omega-3 carboxylic acids) and omega-3-acid ethyl esters (OMACOR®, Abbott Healthcare Products Ltd) following a single oral dose in patients with different degrees of PEI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years and ≤70 years, with suitable veins for cannulation or repeated venipuncture.
* Clinically diagnosed Type 2 diabetics (American Diabetes Association guidelines;), on oral antibiotic drug use ≥3 months and HbA1c value ≥6.5% and ≤9.0% at Visit 1.
* Have a body mass index ≥18 kg/m2 and ≤40 kg/m2 and weigh at least 50 kg.

Exclusion Criteria:

* Intolerance to Omega-3 fatty acids, ethyl esters or fish.
* On insulin therapy or treated with injectable Glucagon-like peptide-1 (GLP-1).
* Treated with bile acid sequestrants.
* Serum levels of TGs >10 mmol/L at any time during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Denmark (3):
  - Research Site, Aarhus
  - Research Site, Frederiksberg
  - Research Site, København NV
- Hungary (3):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Létavértes
- Latvia (3):
  - Research Site, Daugavpils
  - Research Site, Jēkabpils
  - Research Site, Riga
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Puławy
  - Research Site, Staszów
  - Research Site, Zamość
- Slovakia (3):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Ľubochňa
- Sweden (6):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Uppsala

REFERENCES:
- [Derived] Lindkvist B, Nilsson C, Kvarnstrom M, Oscarsson J. Importance of pancreatic exocrine dysfunction in patients with type 2 diabetes: A randomized crossover study. Pancreatology. 2018 Jul;18(5):550-558. doi: 10.1016/j.pan.2018.05.483. Epub 2018 May 19. PMID 29802077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 7 April 2015. Last patient completed Part B: 17 November 2015. This study was performed in 23 centres across 6 countries in Europe.
Pre-assignment Details: A total of 490 patients were screened and of these, 315 patients met all inclusion and none of the exclusion criteria and completed the first part of the study. 51 patients were randomised to treatment in the second part of the study.
Groups:
- Low FEC (EPANOVA® and OMACOR®): Part A investigated serum lipids, especially triglycerides (TGs) and faecal elastase-1 concentration (FEC) as a measure of pancreatic exocrine function in the study population. Patients in the Low FEC group were determined to have FEC levels <100 microgram per gram (mcg/g). No treatment was administered in Part A which was a recruitment phase for Part B. In Part B, study treatment was administered at Visit 4 and Visit 7 with a randomised crossover design to a treatment sequence: AB (a single dose of EPANOVA® 4 g followed by a single dose of OMACOR® 4 g) or BA (a single dose of OMACOR® 4 g followed by a single dose of EPANOVA® 4 g).
- Intermediate FEC (EPANOVA® and OMACOR®): Part A investigated serum lipids, especially TGs and FEC as a measure of pancreatic exocrine function in the study population. Patients in the Intermediate FEC group were determined to have FEC levels ≥100 mcg/g to <200 mcg/g. No treatment was administered in Part A which was a recruitment phase for Part B. In Part B, study treatment was administered at Visit 4 and Visit 7 with a randomised crossover design to a treatment sequence: AB (a single dose of EPANOVA® 4 g followed by a single dose of OMACOR® 4 g) or BA (a single dose of OMACOR® 4 g followed by a single dose of EPANOVA® 4 g).
- Normal FEC (EPANOVA® and OMACOR®): Part A investigated serum lipids, especially TGs and FEC as a measure of pancreatic exocrine function in the study population. Patients in the Normal FEC group were determined to have FEC levels ≥200 mcg/g. No treatment was administered in Part A which was a recruitment phase for Part B. In Part B, study treatment was administered at Visit 4 and Visit 7 with a randomised crossover design to a treatment sequence: AB (a single dose of EPANOVA® 4 g followed by a single dose of OMACOR® 4 g) or BA (a single dose of OMACOR® 4 g followed by a single dose of EPANOVA® 4 g).
Period: Part A (Open-label Recruitment)
Arm/Group | Low FEC (EPANOVA® and OMACOR®) | Intermediate FEC (EPANOVA® and OMACOR®) | Normal FEC (EPANOVA® and OMACOR®)
Started | 16 | 16 | 283
Completed | 16 | 15 | 282
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1
Period: Part B
Arm/Group | Low FEC (EPANOVA® and OMACOR®) | Intermediate FEC (EPANOVA® and OMACOR®) | Normal FEC (EPANOVA® and OMACOR®)
Started | 16 | 15 | 282
Eligible for Randomisation | 15 | 13 | 23
Period 1 Sequence AB | 8 | 6 | 11
Period 1 Sequence BA | 7 | 7 | 12
Period 2 Sequence AB | 8 | 5 | 11
Period 2 Sequence BA | 7 | 7 | 12
Completed | 15 | 12 | 23
Not Completed | 1 | 3 | 259
Not completed — Not randomised to receive treatment | 1 | 2 | 259
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled in Part A that had available serum TG and FEC data (Full Analysis Set) were included in the baseline analysis.
Groups:
- Low FEC (EPANOVA® and OMACOR®): Patients had low levels (<100 mcg/g) of FEC, as determined by the average of the FEC from 2 stool samples collected between Visit 2 and Visit 3 as a measure of pancreatic exocrine function.
- Intermediate FEC (EPANOVA® and OMACOR®): Patients had intermediate levels (≥100 to <200 mcg/g) of FEC, as determined by the average of the FEC from 2 stool samples collected between Visit 2 and Visit 3 as a measure of pancreatic exocrine function.
- Normal FEC (EPANOVA® and OMACOR®): Patients had normal levels (≥200 mcg/g) of FEC, as determined by the average of the FEC from 2 stool samples collected between Visit 2 and Visit 3 as a measure of pancreatic exocrine function.
- Total: Total of all reporting groups
Arm/Group | Low FEC (EPANOVA® and OMACOR®) | Intermediate FEC (EPANOVA® and OMACOR®) | Normal FEC (EPANOVA® and OMACOR®) | Total
Number analyzed (Participants) | 16 | 16 | 283 | 315
Age, Customized [Number; unit: Participants]
  From 18 - 64 years | 11 | 11 | 171 | 193
  From 65 - 84 years | 5 | 5 | 112 | 122
  Over 85 years | 0 | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 5 | 5 | 123 | 133
  Male | 11 | 11 | 160 | 182

OUTCOME MEASURES:

1. Primary Outcome: Part A: Serum TG Level.
Description: For Part A, the distribution of serum TG levels by the degree of pancreatic exocrine insufficiency (PEI) was assessed in patients with Type 2 Diabetes Mellitus (T2DM).
Time Frame: 7 days after enrollment.
Population: The Per Protocol Analysis Set included all enrolled patients without an important protocol deviation.
Measure: Mean (Standard Deviation); unit: millimole per litre (mmol/L)
Groups:
- Low FEC (EPANOVA® and OMACOR®): Part A investigated serum lipids, especially TGs and FEC to assess the relationship between serum TGs and degree of pancreatic exocrine function (as measured by FEC) in the study population. Patients in the Low FEC group were determined to have FEC levels <100 mcg/g. No treatment was administered in Part A which was a recruitment phase for Part B.
- Intermediate FEC (EPANOVA® and OMACOR®): Part A investigated serum lipids, especially TGs and FEC to assess the relationship between serum TGs and degree of pancreatic exocrine function (as measured by FEC) in the study population. Patients in the Intermediate FEC group were determined to have FEC levels ≥100 mcg/g to <200 mcg/g. No treatment was administered in Part A which was a recruitment phase for Part B.
- Normal FEC (EPANOVA® and OMACOR®): Part A investigated serum lipids, especially TGs and FEC to assess the relationship between serum TGs and degree of pancreatic exocrine function (as measured by FEC) in the study population. Patients in the Normal FEC group were determined to have FEC levels ≥200 mcg/g. No treatment was administered in Part A which was a recruitment phase for Part B.
Arm/Group | Low FEC (EPANOVA® and OMACOR®) | Intermediate FEC (EPANOVA® and OMACOR®) | Normal FEC (EPANOVA® and OMACOR®)
Number analyzed (Participants) | 15 | 16 | 278
millimole per litre (mmol/L) | 2.07 (0.63) | 1.68 (0.57) | 2.00 (1.16)

2. Primary Outcome: Part B: Baseline Corrected Area Under the Plasma Concentration Time Curve From Time Zero to Last Measurable Concentration (AUC[0-last]) for Total Eicosapentaenoic Acid (EPA) Following Administration of EPANOVA® and OMACOR®.
Description: Baseline corrected AUC(0-last) was measured for total EPA following administration of single oral doses of EPANOVA® 4 g (A) and OMACOR® 4 g (B) (2-way crossover design) to patients with T2DM and different degrees of PEI.
Time Frame: Blood samples for analysis were taken at 1, 0.5, and 0.05 hours pre-dose, to be used as baseline, and at 1, 2, 3, 4, 5, 6, 7, 8, 10, 24 and 48 hours post-dose.
Population: The Pharmacokinetic (PK) Analysis Set included all randomised patients who received at least one dose of study treatment in Part B and had at least one post-dose PK measurement without any important protocol deviations. 3 subjects were excluded from the analysis for AUC(0-last) due to missing sample results at 48 hours.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*mcg per millilitre (h*mcg/mL)
Groups:
- Low FEC (EPANOVA®); Low FEC (OMACOR®): In Part B, study treatment was administered at Visit 4 (Day 21+5) and Visit 7 (10 to 14 days after Visit 4) with a randomised crossover design. Patients with low FEC, <100 mcg/g were randomised in Part B to a treatment sequence: AB (a single dose of EPANOVA® 4 g followed by a single dose of OMACOR® 4 g) or BA (a single dose of OMACOR® 4 g followed by a single dose of EPANOVA® 4 g).
- Intermediate FEC (EPANOVA®); Intermediate FEC (OMACOR®): In Part B, study treatment was administered at Visit 4 (Day 21+5) and Visit 7 (10 to 14 days after Visit 4) with a randomised crossover design. Patients with intermediate FEC, ≥ 100 to <200 mcg/g, were randomised in Part B to a treatment sequence: AB (a single dose of EPANOVA® 4 g followed by a single dose of OMACOR® 4 g) or BA (a single dose of OMACOR® 4 g followed by a single dose of EPANOVA® 4 g).
- Normal FEC (EPANOVA®); Normal FEC (OMACOR®): In Part B, study treatment was administered at Visit 4 (Day 21+5) and Visit 7 (10 to 14 days after Visit 4) with a randomised crossover design. Patients with normal FEC, ≥ 200 mcg/g, were randomised in Part B to a treatment sequence: AB (a single dose of EPANOVA® 4 g followed by a single dose of OMACOR® 4 g) or BA (a single dose of OMACOR® 4 g followed by a single dose of EPANOVA® 4 g).
Arm/Group | Low FEC (EPANOVA®) | Low FEC (OMACOR®) | Intermediate FEC (EPANOVA®) | Intermediate FEC (OMACOR®) | Normal FEC (EPANOVA®) | Normal FEC (OMACOR®)
Number analyzed (Participants) | 15 | 14 | 13 | 12 | 21 | 22
hours*mcg per millilitre (h*mcg/mL) | 2170 (65.2) | 1650 (31.3) | 2000 (82.8) | 946 (96.0) | 2070 (36.1) | 1260 (126)
Statistical Analysis 1: Comparison: Low FEC (EPANOVA®) vs Low FEC (OMACOR®); Back transformed results are based on the analysis of natural log-transformed data with a Linear Mixed Model containing the terms of FEC classification, treatment, FEC x treatment, sequence, and period as fixed effects and patient nested within sequence as random effect; Test type: Non-Inferiority or Equivalence — The exposure of a single dose of EPANOVA® 4 g (reference) relative to OMACOR® 4 g (test) was estimated by degree of pancreatic exocrine function using level of FEC. Natural log estimates of least-square means (LSmeans) for each treatment and differences of the LSmeans (OMACOR®-EPANOVA®) along with 90% Confidence Intervals (CIs) by degree of pancreatic exocrine function using level of FEC were exponentiated; Geometric least-squares (GLS) Mean Ratio = 0.75, 90% CI 2-sided [0.52 to 1.10] — OMACOR®/EPANOVA®
Statistical Analysis 2: Comparison: Intermediate FEC (EPANOVA®) vs Intermediate FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — The exposure of a single dose of EPANOVA® 4 g (reference) relative to OMACOR® 4 g (test) was estimated by degree of pancreatic exocrine function using level of FEC. Natural log estimates of LSmeans for each treatment and differences of the LSmeans (OMACOR®-EPANOVA®) along with 90% CIs by degree of pancreatic exocrine function using level of FEC were exponentiated; GLS Mean ratio = 0.48, 90% CI 2-sided [0.32 to 0.72] — OMACOR®/EPANOVA®
Statistical Analysis 3: Comparison: Normal FEC (EPANOVA®) vs Normal FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 0.6, 90% CI 2-sided [0.44 to 0.82] — OMACOR®/EPANOVA®

3. Primary Outcome: Part B: Baseline Corrected AUC(0-last) for Total Docosahexaenoic Acid (DHA) Following Administration of EPANOVA® and OMACOR®.
Description: Baseline corrected AUC(0-last) was measured for total DHA following administration of single oral doses of EPANOVA® 4 g (A) and OMACOR® 4 g (B) (2-way crossover design) to patients with T2DM and different degrees of PEI.
Time Frame: as for outcome 2
Population: The PK Analysis Set included all randomised patients who received at least one dose of study treatment in Part B and had at least one post-dose PK measurement without any protocol deviations. 3 subjects were excluded from the analysis for AUC(0-last) due to missing sample results at 48 hours.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Low FEC (EPANOVA®) | Low FEC (OMACOR®) | Intermediate FEC (EPANOVA®) | Intermediate FEC (OMACOR®) | Normal FEC (EPANOVA®) | Normal FEC (OMACOR®)
Number analyzed (Participants) | 15 | 14 | 13 | 12 | 21 | 22
h*mcg/mL | 801 (55.7) | 1040 (47.1) | 719 (85.0) | 567 (70.7) | 625 (90.2) | 810 (105)
Statistical Analysis 1: Comparison: Low FEC (EPANOVA®) vs Low FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 1.28, 90% CI 2-sided [0.84 to 1.93] — OMACOR®/EPANOVA®
Statistical Analysis 2: Comparison: Intermediate FEC (EPANOVA®) vs Intermediate FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 0.80, 90% CI 2-sided [0.51 to 1.25] — OMACOR®/EPANOVA®
Statistical Analysis 3: Comparison: Normal FEC (EPANOVA®) vs Normal FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 1.29, 90% CI 2-sided [0.92 to 1.82] — OMACOR®/EPANOVA®

4. Primary Outcome: Part B: Baseline Corrected AUC(0-last) for Total EPA+DHA Following Administration of EPANOVA® and OMACOR®.
Description: Baseline corrected AUC(0-last) was measured for the sum of EPA and DHA (total EPA+DHA) following administration of single oral doses of EPANOVA® 4 g (A) and OMACOR® 4 g (B) (2-way crossover design) to patients with T2DM and different degrees of PEI.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nanomole/mL (h*nmol/mL)
Arm/Group | Low FEC (EPANOVA®) | Low FEC (OMACOR®) | Intermediate FEC (EPANOVA®) | Intermediate FEC (OMACOR®) | Normal FEC (EPANOVA®) | Normal FEC (OMACOR®)
Number analyzed (Participants) | 15 | 14 | 13 | 12 | 21 | 22
h*nanomole/mL (h*nmol/mL) | 9700 (57.7) | 8780 (32.9) | 8990 (72.4) | 5130 (80.6) | 8890 (43.8) | 6690 (112)
Statistical Analysis 1: Comparison: Low FEC (EPANOVA®) vs Low FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 0.90, 90% CI 2-sided [0.63 to 1.28] — OMACOR®/EPANOVA®
Statistical Analysis 2: Comparison: Intermediate FEC (EPANOVA®) vs Intermediate FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 0.58, 90% CI 2-sided [0.39 to 0.85] — OMACOR®/EPANOVA®
Statistical Analysis 3: Comparison: Normal FEC (EPANOVA®) vs Normal FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 0.75, 90% CI 2-sided [0.55 to 1.00] — OMACOR®/EPANOVA®

5. Primary Outcome: Part B: Baseline Corrected Maximum Plasma Drug Concentration (Cmax) for Total EPA Following Administration of EPANOVA® and OMACOR®.
Description: Baseline corrected Cmax was measured for total EPA following administration of single oral doses of EPANOVA® 4 g (A) and OMACOR® 4 g (B) (2-way crossover design) to patients with T2DM and different degrees of PEI.
Time Frame: as for outcome 2
Population: The PK Analysis Set included all randomised patients who received at least one dose of study treatment in Part B and had at least one post-dose PK measurement without any important protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Low FEC (EPANOVA®) | Low FEC (OMACOR®) | Intermediate FEC (EPANOVA®) | Intermediate FEC (OMACOR®) | Normal FEC (EPANOVA®) | Normal FEC (OMACOR®)
Number analyzed (Participants) | 15 | 15 | 13 | 12 | 22 | 23
mcg/mL | 137 (70.5) | 71.5 (64.0) | 116 (53.3) | 53.9 (70.1) | 131 (36.2) | 69.3 (76.2)
Statistical Analysis 1: Comparison: Low FEC (EPANOVA®) vs Low FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 0.52, 90% CI 2-sided [0.37 to 0.73] — OMACOR®/EPANOVA®
Statistical Analysis 2: Comparison: Intermediate FEC (EPANOVA®) vs Intermediate FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 0.46, 90% CI 2-sided [0.32 to 0.67] — OMACOR®/EPANOVA®
Statistical Analysis 3: Comparison: Normal FEC (EPANOVA®) vs Normal FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 0.53, 90% CI 2-sided [0.40 to 0.70] — OMACOR®/EPANOVA®

6. Primary Outcome: Part B: Baseline Corrected Cmax for Total DHA Following Administration of EPANOVA® and OMACOR®.
Description: Baseline corrected Cmax was measured for total DHA following administration of single oral doses of EPANOVA® 4 g (A) and OMACOR® 4 g (B) (2-way crossover design) to patients with T2DM and different degrees of PEI.
Time Frame: as for outcome 2
Population: The PK Analysis Set included all randomised patients who received at least one dose of study treatment in Part B and had at least one post-dose PK measurement without any protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Low FEC (EPANOVA®) | Low FEC (OMACOR®) | Intermediate FEC (EPANOVA®) | Intermediate FEC (OMACOR®) | Normal FEC (EPANOVA®) | Normal FEC (OMACOR®)
Number analyzed (Participants) | 15 | 15 | 13 | 12 | 22 | 23
mcg/mL | 59.0 (58.6) | 60.5 (47.3) | 56.0 (40.6) | 51.0 (52.0) | 53.8 (41.8) | 59.7 (53.9)
Statistical Analysis 1: Comparison: Low FEC (EPANOVA®) vs Low FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — The exposure of a single dose of EPANOVA® 4 g (reference) relative to OMACOR® 4 g (test) was estimated by degree of pancreatic exocrine function using level of FEC. Natural log estimates of least-squares LSmeans for each treatment and differences of the LSmeans (OMACOR®-EPANOVA®) along with 90% CIs by degree of pancreatic exocrine function using level of FEC were exponentiated; GLS Mean Ratio = 1.02, 90% CI 2-sided [0.77 to 1.36] — OMACOR®/EPANOVA®
Statistical Analysis 2: Comparison: Intermediate FEC (EPANOVA®) vs Intermediate FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS mean Ratio = 0.92, 90% CI 2-sided [0.67 to 1.25] — OMACOR®/EPANOVA®
Statistical Analysis 3: Comparison: Normal FEC (EPANOVA®) vs Normal FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 1.11, 90% CI 2-sided [0.88 to 1.40] — OMACOR®/EPANOVA®

7. Primary Outcome: Part B: Baseline Corrected Cmax for Total EPA+DHA Following Administration of EPANOVA® and OMACOR®.
Description: Baseline corrected Cmax was measured for the sum of EPA and DHA (total EPA+DHA) following administration of single oral doses of EPANOVA® 4 g (A) and OMACOR® 4 g (B) (2-way crossover design) to patients with T2DM and different degrees of PEI.
Time Frame: as for outcome 2
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/mL
Arm/Group | Low FEC (EPANOVA®) | Low FEC (OMACOR®) | Intermediate FEC (EPANOVA®) | Intermediate FEC (OMACOR®) | Normal FEC (EPANOVA®) | Normal FEC (OMACOR®)
Number analyzed (Participants) | 15 | 15 | 13 | 12 | 22 | 23
nmol/mL | 622 (69.7) | 421 (54.0) | 553 (47.0) | 328 (57.2) | 592 (36.6) | 413 (61.7)
Statistical Analysis 1: Comparison: Low FEC (EPANOVA®) vs Low FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean = 0.68, 90% CI 2-sided [0.49 to 0.92] — OMACOR®/EPANOVA®
Statistical Analysis 2: Comparison: Intermediate FEC (EPANOVA®) vs Intermediate FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 0.60, 90% CI 2-sided [0.42 to 0.84] — OMACOR®/EPANOVA®
Statistical Analysis 3: Comparison: Normal FEC (EPANOVA®) vs Normal FEC (OMACOR®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; GLS Mean Ratio = 0.70, 90% CI 2-sided [0.54 to 0.90] — OMACOR®/EPANOVA®

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected until the safety follow-up contact (Visit 10). Serious AEs were collected from Visit 1 (screening) onwards over a period of up to 13 weeks. Other AEs were recorded from Visit 2 over a period of 7 weeks.
Description: Regular investigator assessment at study sites. Population used was the Safety Analysis Set which included all patients who received at least 1 dose of study treatment in Part B.
Groups:
- Low FEC (EPANOVA®): Patients had low levels (<100 mcg/g) of FEC, as determined by the average of the FEC from 2 stool samples collected between Visit 2 and Visit 3 as a measure of pancreatic exocrine function. AEs with an onset date on or after the date of administration of EPANOVA® 4 g at Visit 4 were reported for this group.
- Low FEC (OMACOR®): Patients had low levels (<100 mcg/g) of FEC, as determined by the average of the FEC from 2 stool samples collected between Visit 2 and Visit 3 as a measure of pancreatic exocrine function. AEs with an onset date on or after the date of administration of OMACOR® 4 g at Visit 4 were reported for this group.
- Intermediate FEC (EPANOVA®): Patients had intermediate levels (≥100 to <200 mcg/g) of FEC, as determined by the average of the FEC from 2 stool samples collected between Visit 2 and Visit 3 as a measure of pancreatic exocrine function. AEs with an onset date on or after the date of administration of EPANOVA® 4 g at Visit 4 were reported for this group.
- Intermediate FEC (OMACOR®): Patients had intermediate levels (≥100 to <200 mcg/g) of FEC, as determined by the average of the FEC from 2 stool samples collected between Visit 2 and Visit 3 as a measure of pancreatic exocrine function. AEs with an onset date on or after the date of administration of OMACOR® 4 g at Visit 4 were reported for this group.
- Normal FEC (EPANOVA®): Patients had normal levels (≥200 mcg/g) of FEC, as determined by the average of the FEC from 2 stool samples collected between Visit 2 and Visit 3 as a measure of pancreatic exocrine function. AEs with an onset date on or after the date of administration of EPANOVA® 4 g at Visit 4 were reported for this group.
- Normal FEC (OMACOR®): Patients had normal levels (≥200 mcg/g) of FEC, as determined by the average of the FEC from 2 stool samples collected between Visit 2 and Visit 3 as a measure of pancreatic exocrine function. AEs with an onset date on or after the date of administration of OMACOR® 4 g at Visit 4 were reported for this group.
Arm/Group | Low FEC (EPANOVA®) | Low FEC (OMACOR®) | Intermediate FEC (EPANOVA®) | Intermediate FEC (OMACOR®) | Normal FEC (EPANOVA®) | Normal FEC (OMACOR®)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/13 | 1/12 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 1/15 | 1/15 | 0/13 | 0/12 | 5/23 | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low FEC (EPANOVA®) (N=15) | Low FEC (OMACOR®) (N=15) | Intermediate FEC (EPANOVA®) (N=13) | Intermediate FEC (OMACOR®) (N=12) | Normal FEC (EPANOVA®) (N=23) | Normal FEC (OMACOR®) (N=23)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low FEC (EPANOVA®) (N=15) | Low FEC (OMACOR®) (N=15) | Intermediate FEC (EPANOVA®) (N=13) | Intermediate FEC (OMACOR®) (N=12) | Normal FEC (EPANOVA®) (N=23) | Normal FEC (OMACOR®) (N=23)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Traumatic Ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each Principal Investigator has signed a Confidential Disclosure Agreement which does not allow them to disclose any study related information for 10 years unless it is publically available.